CLINICAL TRIAL: NCT00150852
Title: Vancomycin for Prophylaxis of PEG-Related Wound Infection in MRSA-Positive Patients: a Double-Blind, Randomized, Placebo-Controlled Study
Brief Title: Prevention of Gastrostomy-Related Wound Infection by Vancomycin in Carriers of Methicillin-Resistant Staphylococcus Aureus.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-012 (med 04-008)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2005-09

CONDITIONS: Wound Infection
Keywords: Gastrostomy; Wound infection; Antibiotic prophylaxis
MeSH Terms: conditions — Wound Infection | interventions — Vancomycin

INTERVENTIONS:
Drug: Vancomycin

SUMMARY:
The aim of this study is to determine whether vancomycin with cefazoline is superior to vancomycin with placebo in preventing gastrostomy-related wound infection in carriers of methicillin-resistant staphylococcus aureus (MRSA).

DETAILED DESCRIPTION:
Percutaneous endoscopic gastrostomy (PEG) provides an enteral route for long-term nutrition in patients unable to swallow. Peristomal wound infection occurs in 5 - 30 % of patients. Systematic antibiotic prophylaxis by cephalosporins or ampicillin/clavulanic acid has been shown to prevent this complication efficiently.

MRSA-positive patients have been suggested to be at higher risk of PEG-related wound infection due to MRSA. However, recommendations about vancomycin-prophylaxis before surgical procedures have not been extended to PEG insertion. This might be due to the fact that the exact route of contamination is unknown. It is assumed that contamination occurs when gastrostomy tubes are passed through the oropharynx. However, oropharyngeal carriage appears less frequent than nasopharyngeal or cutaneous carriage. Furthermore, patients who receive PEG are particularly vulnerable to vancomycin toxicity because of older age and multiple comorbidities.

The aim of this study is to compare the rate of infectious complications after PEG insertion in patients colonized with MRSA who received either standard intravenous antibiotic prophylaxis associated with vancomycin or standard prophylaxis with placebo.

ELIGIBILITY:
Inclusion Criteria:

* PEG insertion in a patient with a swab positive for MRSA during the 4 weeks preceding PEG insertion

Exclusion Criteria:

* Age < 18 years
* No informed consent obtained either from the patient or from his legal representative
* Contraindication to the administration of cefazolin or of vancomycin
* Systemic administration of antibiotics effective against MRSA during the week prior to the procedure
* Technique of PEG insertion different from the standard pull technique proposed by the physician in charge and the gastroenterologist
* Patients requiring antibiotic prophylaxis of endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Start 2004-09

PRIMARY OUTCOMES:
Rate of PEG-site infection at 3, 7, 14, 21 and 28 days post intervention as assessed by a clinical score (Jain score) and swab culture

SECONDARY OUTCOMES:
Additional costs and nursing charges (Programme de Recherche en Nursing (PRN) scoring system)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Vonlaufen, MD, Principal Investigator — Division of Gastroenterology, University Hospital, Geneva
Locations (3):
- Centre Hospitalier Universitaire (CHU), Grenoble, France
- Switzerland (2):
  - Division of Gastroenterology, University Hospital, Geneva, Canton of Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud